CLINICAL TRIAL: NCT05143463
Title: A Phase 1, Randomized, Placebo-controlled, Double-blind, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous NS101 Infusion in Healthy Volunteers
Brief Title: A FIH Study to Assess the Safety and Tolerability of NS Intravenous NS101 Infusion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuracle Science Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NS101_P1_01
Record Dates: First submitted 2021-10-29; First posted 2021-12-03 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Neurodegenerative Diseases
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Intervention Model Description: For each dose level, the dose to be administered to each subject for a single infusion will be calculated based on subject's body weight, measured on Day 1.
Who Masked: Participant, Investigator
Masking Description: Subjects will be administered each treatment (NS101 or placebo), according to the block randomization scheme. The subjects and the clinical personnel involved in the collection, monitoring, revision, or evaluation of AEs, or personnel who could have an impact on the outcome of the study will be blinded with respect to the subject's treatment assignment (NS101 or placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential SAD - NS101 (Experimental): A staggered dosing schedule will be used for each dose level administered under fasting conditions.
  Interventions: Drug: NS101 IV infusion
- Sequential SAD - NS101 Placebo (Placebo Comparator): Volume of matching placebo will be determined based on subject weight and NS101 concentration per cohort.
  Interventions: Drug: NS101 IV infusion

INTERVENTIONS:
Drug: NS101 IV infusion — Approximately 1 hour prior to start of study drug infusion, an IV port will be inserted into the antecubital region and a sterile normal saline solution infusion will be initiated at fixed rate in order to keep the vein open. The study drug will be infused over approximately 60 minutes at a constant rate. At the end of the infusion, 3 mL of saline solution will be injected to flush the remaining drug into the IV catheter. The end of infusion will be set to the end of the 3 mL flush. For safety reason (e.g., administration of rescue medication), the IV line will remain opened for approximately 1 hour following completion of infusion.

SUMMARY:
Up to 80 healthy adult males, ≥ 18 and ≤ 55 years of age, are planned to be enrolled in the study.

The study will consist of 8 cohorts (Cohorts 1 to 8, 1 cohort per dose level). Each cohort will include 8 subjects (6 subjects receiving a single dose of the study drug NS101 and 2 subjects receiving a single dose of a matching placebo), for a total of 64 subjects planned for evaluation. A total of 21 blood samples will be collected in each cohort for PK analysis and a total of 14 blood samples will be collected in each cohort for PD analysis.

DETAILED DESCRIPTION:
The study will consist of 8 cohorts (Cohorts 1 to 8, 1 cohort per dose level). Each cohort will include 8 subjects (6 subjects receiving a single dose of the study drug NS101 and 2 subjects receiving a single dose of a matching placebo), for a total of 64 subjects planned for evaluation.

For each dose level, the dose to be administered to each subject for a single infusion will be calculated based on subject's body weight, measured on Day 1.

In each cohort, subjects will receive a single infusion of NS101 or matching placebo under fasting conditions over a period of approximately 60 minutes at the target dose level. A total of 21 blood samples will be collected in each cohort for PK analysis and a total of 14 blood samples will be collected in each cohort for PD analysis. A total of 6 immunogenicity blood samples will be collected for ADA and NAbs. For each subject in cohort 5 to 8 only, one single CSF sample will be collected via lumbar puncture over the study, for PK and PD analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male, non-smokers (no use of tobacco or nicotine products within 6 months prior to screening), ≥18 and ≤55 years of age, with BMI >18.5 and <30.0 kg/m2 and body weight ≥50.0 kg for males.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to dosing.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Subject's score on the Sheehan Suicidality Tracking Scale (S-STS) at screening must be 0.

Exclusion Criteria:

1. Any clinically significant abnormality at physical examination, clinically significant abnormal laboratory test results or positive test for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C found during medical screening.
2. Positive urine drug screen or alcohol breath test at screening or admission.
3. History of asthma, allergic rhinitis or urticaria, anaphylactic reactions, or any other clinically significant allergic reactions to any medication, including biologics, or food, or allergy to any excipient in the formulation.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
AEs of NS101 following intravenous (IV) administration of single ascending doses in healthy subjects | up to 60 Days ± 3 after IV infusion
  To assess Incidence, nature, relatedness, and severity of adverse events (AEs) of NS101 following intravenous (IV) administration of single ascending doses in healthy subjects

SECONDARY OUTCOMES:
AUC of NS101 in serum | up to 1416 hours after IV infusion
  To characterize the pharmacokinetic (PK) profile of NS101 in serum following single IV infusion doses in healthy subjects
Cmax of NS101 in serum | up to 1416 hours after IV infusion
  To characterize the pharmacokinetic (PK) profile of NS101 in serum following single IV infusion doses in healthy subjects
Concentrations of FAM19A5 in Cerebrospinal fluid (CSF) | up to 336 hours after IV infusion
  To investigate FAM19A5 concentrations in CSF following single IV infusion doses in healthy subjects for Cohort 5 to 8 only
The immunogenicity profile of NS101 | up to 1416 hours after IV infusion
  To measure as the number and percentage of subjects who develop detectable Anti-Drug Antibody (ADA) and Neutralizing Antibody (NAb).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, M.D., Principal Investigator — Syneos Health
Locations (1):
- Syneos Health, Québec, Canada

IPD SHARING:
Plan to Share IPD: No
Will decide once CSR is released

REFERENCES:
- [Derived] Kim HB, Yoo S, Kwak H, Ma SX, Kim R, Lee M, Ha N, Pyo S, Kwon SG, Cho EH, Lee SM, Jang J, Kim WK, Park HC, Baek M, Park Y, Park JY, Park JW, Hwang SW, Hwang JI, Seong JY. Inhibition of FAM19A5 reverses synaptic loss and cognitive decline in mouse models of Alzheimer's disease. Alzheimers Res Ther. 2025 Jul 21;17(1):168. doi: 10.1186/s13195-025-01813-8. PMID 40691577

DOCUMENTS (2):
  • Study Protocol (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT05143463/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT05143463/SAP_001.pdf